CLINICAL TRIAL: NCT05468385
Title: Transcutaneous Auricular Vagus Nerve Stimulation Improves Inhibitory Control in Emotional Go-Nogo Task
Brief Title: The Effects of taVNS on Inhibitory Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UESTC-neuSCAN-90
Record Dates: First submitted 2022-07-15; First posted 2022-07-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tragus stimulation (Experimental): Vagus nerve stimulation via tragus
  Interventions: Device: Vagus nerve stimulation via tragus
- Sham stimulation (Sham Comparator): Sham stimulation via earlobe
  Interventions: Device: Sham stimulation via earlobe

INTERVENTIONS:
Device: Vagus nerve stimulation via tragus — The device will send stimulus intensity of around 0.5mA via tragus in the left ear (based on participants' subjective report), delivered with a pulse width of 0.5 ms at 25 Hz. Stimulation will be active for 30 seconds, followed by a break of 30 seconds.
  Arms: Tragus stimulation
Device: Sham stimulation via earlobe — The device will send stimulus intensity of around 0.5mA via the earlobe in the left ear (based on participants' subjective reports), delivered with a pulse width of 0.5 ms at 25 Hz. Stimulation will be active for 30 seconds, followed by a break of 30 seconds.
  Arms: Sham stimulation

SUMMARY:
The main aim of the study is to investigate whether the transcutaneous vagus nerve stimulation(tVNS) improves the ability of inhibitory control in an emotional Go-Nogo task.

DETAILED DESCRIPTION:
A randomized, sham-controlled, between-subject design will be employed in this study. A total of 87 healthy subjects will receive either transcutaneous vagus nerve stimulation via tragus or sham stimulation via the earlobe in the left ear. Brain activity and behavioral data for an emotional Go-Nogo task will be recorded and saliva samples will be collected before, during, and after stimulation.

Some personal traits will be assessed using different kinds of questionnaires, such as the State-Trait Anxiety Inventory (STAI), Beck's Depression Inventory(BDI), Autism Spectrum Quotient (ASQ) et al.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* pregnant, menstruating, taking oral contraceptives;
* medical or psychiatric illness.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
The ability of inhibitory control in an emotional Go-Nogo task | After 30 minutes stimulation
  Analysis the behavioral and brain data recorded during the task
Oxytocin release | within 5 minutes after taVNS via tragus and earlobe
  Investigating the oxytocin release after taVNS via tragus and earlobe based on saliva samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No